CLINICAL TRIAL: NCT01465243
Title: An Open , Single-Center, Single Arm Trial to Evaluate the Efficacy and Safety of Dose Escalation of Icotinib in Advanced NSCLC Patients After Routine Icotinib Therapy
Brief Title: Dose Escalation Of Icotinib In Previously Treated Patients With Routine Dose
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-IC-IV01
Record Dates: First submitted 2011-11-01; First posted 2011-11-04 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Efficacy; Safety; EGFR-TKI; phase IV; NSCLC; Dose escalation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Icotinib (Experimental): This is a single arm study.
  Interventions: Drug: Icotinib

INTERVENTIONS:
Drug: Icotinib — 125 mg Tid (375 mg per day) 250 mg Tid (750 mg per day)
  Other Names: BPI-2009, Conmana

SUMMARY:
To determine whether dose escalation can provide a better survival to patients who failed with icotinib at routine dose.

DETAILED DESCRIPTION:
Lung cancer is a major cause of morbidity and mortality, which is the rapidest increased type of cancer in China with over 5 times incidence rate increase during the past 30 years. Tyrosine kinase inhibitors (TKIs) of the epidermal growth factor receptor (EGFR) have been widely used for the treatment of patients with non-small cell lung cancer(NSCLC). Icotinib is a novel EGFR-TKI developed by a group of Chinese scientists and clinician. Icotinib appears to be non-inferior to Gefitinib in terms of efficacy, better in terms of safety, and larger of therapeutic window in phase I-III trials. In this study, an open , single-center, single arm phase IV trial was designed to evaluate the safety and efficacy of dose escalation of icotinib in the treatment of advanced NSCLC patients after failure with routine dose. PFS (progress free survival) is the primary end-point with OS (overall survival), ORR (objective response), TTP (time to progress), HRQOL and safety as the secondary end-point.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed NSCLC with Histology or cytology; advanced （IIIb/IV).
2. Must have received 1 or 2 chemotherapy (at least 1 is platin based)before, and prior chemotherapy must be completed at least 4 weeks before study enrollment.
3. Measurable, evaluable disease outside of a radiation port.

Exclusion Criteria:

1. Previous usage of EGFR-TKI or antibody to EGFR: gefitinib, erlotinib, herceptin, erbitux.
2. Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-09; Primary Completion 2013-10 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Progression-free Survival | 6-12 months

SECONDARY OUTCOMES:
Overall survival | 6 months -1 year
Objective response rate | 3-6 months
Time to progression | 3-6 months
Health-Related Quality of Life (HR QOL) | 1 year
Number of Participants with adverse events and serious adverse events (SAEs) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Li Xi qing, M.D., Principal Investigator — 307 Hospital of People's Liberation Army（PLA）
Locations (1):
- 307 Hospital of People's Liberation Army（PLA）, Beijing, Beijing Municipality, China